CLINICAL TRIAL: NCT01314040
Title: Study to Identify Biomarkers for Protein Intake; a Randomized, Fully Controlled Feeding Study
Brief Title: Study to Identify Biomarkers for Protein Intake
Acronym: Biomarker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: J.M. Geleijnse PhD, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A1003/ WP-B1
Record Dates: First submitted 2011-02-25; First posted 2011-03-14 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Identify New Biomarkers in Blood or Urine After Consumption of Meat Protein, Dairy Protein and Grain Protein in Healthy Subjects.
Keywords: Dietary protein; Biomarkers; filtration rate; urinary acid excretion
MeSH Terms: interventions — Jogging; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Run in (Other)
  Interventions: Other: Run in diet
- High meat protein diet (Experimental)
  Interventions: Other: High meat protein diet
- High dairy protein diet (Experimental)
  Interventions: Other: High dairy protein diet
- High grain protein diet (Experimental)
  Interventions: Other: High grain protein diet

INTERVENTIONS:
Other: Run in diet — Fully controlled dietary period during 9 days. Participants will receive approximately 15 en% of protein. The amount of protein intake from dairy, meat, and grain will be equal to each other
  Arms: Run in
Other: High meat protein diet — Fully controlled diet during 7 days. Participants will consume 18 en% protein, mainly from meat.
  Arms: High meat protein diet
Other: High dairy protein diet — Fully controlled dietary intervention during 7 days. Participants will consume 20 en% protein. Mainly from dairy
  Arms: High dairy protein diet
Other: High grain protein diet — Fully controlled dietary intervention for 7 days. Participants will consume 20 en% of protein. Mainly from grain
  Arms: High grain protein diet

SUMMARY:
Results from observational studies suggest a small beneficial association between protein and blood pressure that may be mainly attributable to the intake of protein from plant sources. In epidemiological studies biomarkers of dietary intake are useful to estimate intake more reliably. Dietary studies using biomarkers of protein intake generally show stronger associations with health outcomes. However, data on biomarkers for specific types of protein (e.g. from dairy, meat, grain and legumes) are scarce. Therefore the purpose of this study is to identify new biomarkers for the intake of protein from meat, dairy and grain. In addition the secondary purpose is to investigate whether intake of protein from these sources influences kidney filtration rate and urinary acid excretion differentially.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* BMI between 18.5 and 30 kg/m2
* Healthy (As judged by the participant)
* Written informed consent obtained

Exclusion Criteria:

* Unable or unwilling to comply with study procedures.
* Unusual dietary patterns, including high alcohol intakes (≥ 2 glasses/day) and a vegetarian diet
* Recent (< 4 weeks) or current participation in a study with any investigational drug or dietary intervention
* Usage of an energy restricted diet during the last two months
* Weight loss or weight gain of 5 kg or more during the last two months
* Smoking
* Stomach or bowel diseases
* Kidney disorders
* Diabetes, thyroid disease, other endocrine disorders
* Prevalent cardiovascular disease
* Extreme sports (>8h/ wk)
* Usage of any prescribed medication except for oral contraceptives
* Use of systemic antibiotics in the period of 3 month prior to the study
* For women: pregnant or lactating
* For women: not using oral contraceptives
* For women: Unwilling to use oral contraceptives for consecutively for at least the total study duration
* Liver function parameters (ALAT, ASAT, and γ-GT) and renal function parameters (Serum creatinin) outside the normal range

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Differences between dietary periods in concentrations of potential biomerkers in blood and urine | On the last day of every one week intervention period
  Potential biomarkers that will be measured are urinary creatinin, sulphate, carnosine, 1-MH, 3-MH, taurine,14N/15N and creatin in blood. Furthermore, amino acid profiling will be done in blood and urine to detect differences between dietary periods

SECONDARY OUTCOMES:
Differences between dietary period in estimated renal filtration | blood and urine collection on the last day of each intervention period
  Renal filtration will be estimated using bromide distribution in combination with bio-impedance measurement
Differences between dietary periods in urinary acid excretion | urine collection on the last day of each intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

REFERENCES:
- [Derived] Vissers LET, Soedamah-Muthu SS, van der Schouw YT, Zuithoff NPA, Geleijnse JM, Sluijs I. Consumption of a diet high in dairy leads to higher 15:0 in cholesteryl esters of healthy people when compared to diets high in meat and grain. Nutr Metab Cardiovasc Dis. 2020 May 7;30(5):804-809. doi: 10.1016/j.numecd.2020.01.006. Epub 2020 Jan 25. PMID 32139254